CLINICAL TRIAL: NCT01614821
Title: Phase 2 Study of Bruton's Tyrosine Kinase (Btk) Inhibitor, Ibrutinib (PCI-32765), in Waldenstrom's Macroglobulinemia
Brief Title: Ibrutinib (PCI-32765) in Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Steven P. Treon, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-015
Record Dates: First submitted 2012-05-17; First posted 2012-06-08 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Recurrence | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): PCI-32765; ibrutinib
  Interventions: Drug: PCI-32765

INTERVENTIONS:
Drug: PCI-32765 — Taken orally, once daily in the morning
  Other Names: ibrutinib

SUMMARY:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational drug, PCI-32765, to learn whether PCI-32765 works in treating a specific cancer. "Investigational" means that PCI-32765 is still being studied and that research doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause, and if PCI-32765 is effective for treating different types of cancer. It also means that the FDA has not yet approved PCI-32765 for use in patients, including people with Waldenstrom's Macroglobulinemia.

PCI-32765 is a newly discovered drug that is being developed as an anti-cancer agent. PCI-32765 is a Bruton's tyrosine kinase (Btk) inhibitor drug which interrupts B cell receptor (BCR) signaling in lymphomas by selectively and irreversibly binding to the Btk protein, which then results in malignant cell death. This drug has been used in laboratory experiments and other research studies in B-cell malignancies and information from those other research studies suggests that PCI-32765 may be a treatment strategy for B-cell malignancies, including Waldenstrom's Macroglobulinemia.

In this research study, the investigators are testing the safety and efficacy of PCI-32765 as a treatment option for relapsed or refractory Waldenstrom's Macroglobulinemia.

DETAILED DESCRIPTION:
Patients in this research study will receive up to 40 cycles of treatment. Each treatment cycle lasts 4 weeks. Patients will take PCI-32765 by mouth, once a day in the morning.

During each cycle patients will be asked to visit the clinic for scheduled tests and exams and to receive a supply of PCI-32765 to take at home every day. Patients will visit the clinic on the first day of each of the first 3 cycles, and then just once at the beginning of every three cycles.

During study visits, patients will have a physical exam where they will be asked questions about their general health and specific questions about any problems that they might be having and any medications they may be taking. Patients will have blood tests to see how their disease is responding to the study treatment and how they are tolerating the study drug. Patients may also have CT scans of the chest, abdomen and pelvis as well as a bone marrow aspirate and biopsy. If a patient's disease stays the same or is helped, he/she will continue to get study treatment. If disease worsens, he/she will be taken off study treatment at that time.

After completion of the treatment and as part of standard of care, follow-up tests will include a physical exam, review of symptoms and medications, blood tests, bone marrow aspirate and biopsy, CT scans of the chest, abdomen and pelvis. The investigators would like to continue to monitor progress by following-up every three months for up to two years after completion of study treatment or until next treatment, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenstrom's Macroglobulinemia
* Measurable disease
* Have received at least one prior therapy for WM therapies
* Disease free of prior malignancies
* Able to adhere to study visit schedule and other protocol requirement

Exclusion Criteria:

* Pregnant or breastfeeding
* Any other serious medical condition
* Concurrent use of other anti-cancer agents or treatments
* Prior exposure to PCI-32765
* Known CNS lymphoma
* Significant cardiovascular disease
* Any disease affecting gastrointestinal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2018-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Treon, MD PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Guijosa A, Ramirez-Gamero A, Sarosiek S, Branagan AR, von Keudell G, Treon SP, Castillo JJ. Ibrutinib plus rituximab vs ibrutinib monotherapy in patients with Waldenstrom macroglobulinemia: a pooled analysis. Blood Adv. 2025 Sep 23;9(18):4705-4715. doi: 10.1182/bloodadvances.2025016536. PMID 40674744
- [Derived] Treon SP, Meid K, Gustine J, Yang G, Xu L, Liu X, Patterson CJ, Hunter ZR, Branagan AR, Laubach JP, Ghobrial IM, Palomba ML, Advani R, Castillo JJ. Long-Term Follow-Up of Ibrutinib Monotherapy in Symptomatic, Previously Treated Patients With Waldenstrom Macroglobulinemia. J Clin Oncol. 2021 Feb 20;39(6):565-575. doi: 10.1200/JCO.20.00555. Epub 2020 Sep 15. PMID 32931398
- [Derived] Treon SP, Tripsas CK, Meid K, Warren D, Varma G, Green R, Argyropoulos KV, Yang G, Cao Y, Xu L, Patterson CJ, Rodig S, Zehnder JL, Aster JC, Harris NL, Kanan S, Ghobrial I, Castillo JJ, Laubach JP, Hunter ZR, Salman Z, Li J, Cheng M, Clow F, Graef T, Palomba ML, Advani RH. Ibrutinib in previously treated Waldenstrom's macroglobulinemia. N Engl J Med. 2015 Apr 9;372(15):1430-40. doi: 10.1056/NEJMoa1501548. PMID 25853747

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 63
Completed | 63
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 31
Age, Continuous [Median (Standard Deviation); unit: years] | 63 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To assess the overall response rate (>25% reduction in serum IgM from baseline).
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 63
Participants | 57

2. Secondary Outcome: Safety and Tolerability of PCI-32765
Description: To assess the safety and tolerability of PCI-32765 in symptomatic WM patients with relapsed/refractory disease. Grade > or = 2 Adverse Events determined to be associated with PCI-32765 and subsequent outcomes will constitute the safety profile of PCI-32765 in WM. Percent of participants who experienced at least 1 grade 2 or higher treatment emergent adverse event.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 63
Participants | 62

3. Secondary Outcome: Determine Progression Free Survival
Description: To determine Progression Free Survival (PFS in symptomatic WM patients with relapsed/refractory disease. Participants were treated for 40 cycles and then followed for 2 years or until next therapy or death. 40 participants were censored prior to disease progression.
Time Frame: 6 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 63
months | 39 [0 to 67]

4. Secondary Outcome: To Determine Time to Next Therapy (TTNT) of PCI-32765 in Symptomatic WM Patients With Relapsed/Refractory Disease
Description: Time to Next Therapy is the duration of time from of starting ibrutinib until next therapy. Participants were treated for 40 cycles and then followed for 2 years or until next therapy or death. Participants had the option to continue ibrutinib commercially. 40 participants were censored while still on commercial ibrutinib therapy.
Time Frame: 6 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 63
months | 49 [1 to 67]

5. Secondary Outcome: Major Response Rates
Description: To assess the major response rate (>50% reduction in serum IgM from baseline)
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 63
Participants | 49

6. Secondary Outcome: Very Good Partial Response Rate
Description: To assess the very good partial response rate (>90% reduction in serum IgM from baseline)
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 63
Participants | 17

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Cycle 1 Day 1 through 30 days after discontinuing protocol ibrutinib therapy, an average of 3 years.
Description: Grade 2 and above treatment emergent adverse events were collected.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 1/63
Serious Adverse Events (participants affected / at risk) | 30/63
Other Adverse Events (participants affected / at risk) | 62/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=63)
Fever and Tachycardia (General disorders) | 1 (1)
Flu (Infections and infestations) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Neutropenic Fever and Chills (Blood and lymphatic system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Malaise (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 11 (11)
Endocarditis (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Disease Transformation DLBCL (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Group A Streptococcus (Infections and infestations) | 1 (1)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Platelet Count Decreased (Investigations) | 2 (2)
Neutrophil count Decreased (Investigations) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1)
Adenocarcinoma of the rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Depression and Suicidal Ideation (Psychiatric disorders) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Foot Infection (Infections and infestations) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=63)
Abdominal Pain (Gastrointestinal disorders) | 7 (7)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 40 (40)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (17)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Bladder Infection (Infections and infestations) | 3 (3)
Bloating (Gastrointestinal disorders) | 3 (3)
Blood bilirubin increased (Investigations) | 4 (4)
Blurred vision (Eye disorders) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bronchial infection (Infections and infestations) | 7
Bruising (Injury, poisoning and procedural complications) | 8 (8)
Cataract (Eye disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 3 (3)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Depression (Psychiatric disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 20 (20)
Dizziness (Nervous system disorders) | 11 (11)
Dry eye (Skin and subcutaneous tissue disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Facial edema (General disorders) | 1 (1)
Edema limbs (General disorders) | 9 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Eye infection (Infections and infestations) | 1 (1)
Eye pain (Eye disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 33 (33)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 13 (13)
Fly-like symptoms (General disorders) | 4 (4)
Fracture (Injury, poisoning and procedural complications) | 4 (4)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 12 (12)
Gum infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 11 (11)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hematoma (Vascular disorders) | 5 (5)
Hematuria (Renal and urinary disorders) | 4 (4)
Hemorrhoidal hemmorhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 9 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Lipase increased (Investigations) | 2 (2)
Lung infection (Infections and infestations) | 14 (14)
Lymphedema (Vascular disorders) | 1 (1)
Malaise (General disorders) | 6 (6)
Mucosal infection (Infections and infestations) | 3 (3)
Oral Mucositis (Gastrointestinal disorders) | 8 (8)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (14)
Nail infection (Infections and infestations) | 3 (3)
Nail ridging (Skin and subcutaneous tissue disorders) | 7 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 9 (9)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 26 (26)
Non-cardiac chest pain (General disorders) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 4 (4)
Otitis media (Infections and infestations) | 3 (3)
Pain (General disorders) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Palpiatations (Cardiac disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 7 (7)
Penile Infection (Infections and infestations) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 9 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (12)
Pharyngitis (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 29 (29)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 5 (5)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (7)
Rectal perforation (Gastrointestinal disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Retinal detachment (Eye disorders) | 2 (2)
Retinal tear (Eye disorders) | 1 (1)
scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Sinusitis (Infections and infestations) | 21 (21)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 11 (11)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tinnitis (Ear and labyrinth disorders) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 19 (19)
Urinary tract infection (Infections and infestations) | 9 (9)
urinary tract obstruction (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Vaginal infection (Infections and infestations) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7)
Watering eyes (Eye disorders) | 1 (1)
Weight gain (Investigations) | 2 (2)
Weight loss (Investigations) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No